CLINICAL TRIAL: NCT00000126
Title: Ischemic Optic Neuropathy Decompression Trial Followup (IONDT Followup)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Other Study IDs: NEI-25
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2003-10

CONDITIONS: Ischemic Optic Neuropathy
Keywords: Non-arteritic Ischemic Optic Neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Procedure: Surgery

SUMMARY:
To follow all patients enrolled in the original Ischemic Optic Neuropathy Decompression Trial (IONDT) to determine (1) the incidence of non-arteritic ischemic optic neuropathy (NAION) in the second eye, (2) changes in visual acuity over time in both the study and second eye, and (3) other aspects of the natural history of NAION.

DETAILED DESCRIPTION:
NAION is the most common cause of acute optic nerve disease in the elderly, causing permanent and severe visual loss. No proven treatment currently exists to reverse or arrest this loss. There is no accepted method for the prevention or reduction of the likelihood of second eye involvement. NAION strikes both eyes in as many as 40 percent of affected patients (Beri et al. 1987), with a 2-year risk of about 25 percent (Steven Feldon, personal communication to SEK).

IONDT compared optic nerve decompression surgery (ONDS), which was becoming a widely used treatment for NAION, with careful followup alone, in patients with newly diagnosed NAION. The rationale for the surgery was that NAION was caused by impaired blood flow to the optic nerve and that decompression surgery would restore vision by alleviating pressure surrounding the nerve. Because ONDS was fast becoming the standard of care, evaluation of the safety and efficacy of the procedure was tested in the context of a randomized clinical trial.

Within 2 years of the start of the IONDT, the Data and Safety Monitoring Committee recommended cessation of the clinical trial recruitment. The National Institutes of Health issued a clinical alert to 25,000 ophthalmologists and neurologists describing the study findings that surgery was no better than careful followup and may be harmful (IONDT 1995). It was recommended that ONDS not be used in cases of NAION. Thus, the IONDT findings not only have led to a costly and ineffective surgery to be abandoned as a treatment for NAION, but also have left practitioners with a dearth of treatment choices.

The IONDT is the first multicenter, prospective study of newly diagnosed patients with NAION. The baseline history and examination, which took place within 14 days of the onset of symptoms, used standardized methods and diagnostic criteria to collect data on all factors possibly relating to the etiology of NAION. In reports from previous studies that present data on both initial and final visual acuities, no data are available regarding change in visual acuity over time for individual patients. Where data are available on final visual acuity, reported rates of improvement are low, ranging from 0 percent to 33 percent for untreated eyes. The IONDT found, however, an improvement of three or more lines in 42.7 percent of patients who received careful followup.

NAION in both eyes has been reported in as few as 10.5 percent and as many as 73 percent of patients. In a study of bilateral NAION where all patients were prospectively logged, Beri et al. reported that 17.5 percent of patients developed bilateral disease at 1 year of followup and 34.5 percent developed it at 5 years. However, Beck et al., using a life table analysis on the same cohort reported by Beri et al., estimated the risk of bilateral NAION to be 12 percent within 2 years and 19 percent within 5 years. The IONDT has so far similarly reported a 12 percent (25/216) incidence of bilateral NAION in its randomized patients. The incidence in the nonrandomized group, 91 percent of whom had visual acuity better than 20/64, is much lower at 4 percent (5/136).

Thus, continued followup of the IONDT cohort is critically important to ascertain a clear picture of the natural history of NAION in terms of involvement of the second eye and long-term vision. Data obtained will be critical in understanding the etiology of the disease and in generating hypotheses for testing further treatments for the disease.

The IONDT Followup Study will continue to monitor vision and other health outcomes in patients originally enrolled in the IONDT, whether randomized to one of the two treatment groups or whether followed as part of the natural history cohort. All IONDT patients were diagnosed with NAION within 14 days of onset of symptoms, have had a minimum of 2 years of continuous followup, and will be followed for an additional 4 years in the Followup Study. Patients will have annual visits at the original IONDT Clinical Center or, if necessary, with a surrogate provider. If NAION occurs in the second eye, the patient will be asked to visit the clinic for a special visit. The Coordinating Center will telephone the patients on a quarterly basis, between annual visits. Outcomes that will be examined include:

* incidence of NAION in the second eye,
* medical or ocular events surrounding the occurrence of NAION,
* visual acuity (measured using the New York Lighthouse charts).

In the event of an NAION event in the second eye, the patient's visual field will be tested by using the Humphrey Perimeter.

ELIGIBILITY:
All living patients from the 420 patients originally enrolled in the IONDT have been asked to participate in the IONDT Followup Study. No new patients are being recruited.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-10

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Doheny Eye Institute, University of Southern California, Los Angeles, California
  - Jules Stein Eye Institute, Los Angeles, California
  - Department of Ophthalmology, University of California, San Francisco, San Francisco, California
  - Department of Ophthalmology, University of Florida, Gainesville, Florida
  - Emory Eye Center, Emory University, Atlanta, Georgia
  - Department of Ophthalmology, University of Illinois, Chicago, Illinois
  - Department of Ophthalmology, University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - W.K. Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Department of Ophthalmology, Michigan State University, East Lansing, Michigan
  - William Beaumont Eye Institute, William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mason Institute of Ophthalmology, University of Missouri - Columbia, Columbia, Missouri
  - St. Louis University, Anheuser-Busch Eye Institute, St Louis, Missouri
  - SUNY Health Science Center, Department of Neurology, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of South Carolina, Department of Ophthalmology, Columbia, South Carolina
  - University of Texas, Houston, Texas
  - University of Utah, Department of Ophthalmology, Salt Lake City, Utah
  - University of Virginia, Department of Ophthalmology, Charlottesville, Virginia
  - Medical College of Virginia, Department of Neurology, Richmond, Virginia
  - West Virginia University, Department of Neurology, Morgantown, West Virginia